CLINICAL TRIAL: NCT05354817
Title: Re-Play: Impact of FOLFIRINOX Chemotherapy in IV Colorectal Cancer Patients Previously Exposed to Irinotecan, Fluoropyrimidine and Oxaliplatin
Brief Title: Impact of FOLFIRINOX Chemotherapy in IV Stage Colorectal Cancer Patients Previously Exposed to Irinotecan, Fluoropyrimidine and Oxaliplatin
Acronym: Re-Play
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 1950
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer Stage IV
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mFolfirinox (Other)
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: mFOLFIRINOX — mFOLFIRINOX: - Oxaliplatin; Leucovorin; Irinotecan and 5-FU

SUMMARY:
The purpose of this work is to verify prospectively what the rate of response after triple chemotherapy with mFOLFIRINOX in patients in IV stage of Colorectal Cancer who have already failed after at least two lines of dual combinations with fluoropyrimidine, oxaliplatin, irinotecan and anti-EGFR if wild-type RAS.

Currently at ICESP, patients are frequently re-exposed in third line to double combinations.

DETAILED DESCRIPTION:
Single-arm phase II study. The chemotherapy regimen with mFOLFIRINOX will be administered every 14 for 4 cycles, after evaluation of tumor response, you can maintain treatment until disease progression.

The FOLFIRINOX regimen, as well as the drugs used (oxaliplatin, 5-Fluorouracil, leucovorin and irinotecan) is already indicated in the package insert for the treatment of colorectal cancer.

If treatment is discontinued after cycle 4 with the patient responding, for response maximum or unmanageable toxicity, it is suggested to maintain imaging control every 60 days (7-day window) until disease progression. This interval is already commonly used for patients with metastatic disease who are on treatment pause. Treatment in progression of illness will be at the discretion of the treating physician. Cancer patients undergoing chemotherapy routinely perform evaluation of organ functions and CEA, as well as clinical evaluation before each cycle of treatment

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic colon/rectal adenocarcinoma, with measurable by RECIST v. 1.1
* Disease progression to at least two lines of chemotherapy with chemotherapy regimens that contain fluoropyrimidine, irinotecan and oxaliplatin
* Patients with RAS research in tumor sample with result wild animals must have previously received anti-EFGR therapy.
* ECOG (Eastern Cooperative Oncology Group) 0 or 1
* Availability of tumor material for molecular analysis
* Hb > 8, neutrophils > 1,500 and PLQ > 100,000
* Adequate kidney and liver function

Exclusion Criteria:

* Active neoplasm with other primary site, except in situ tumors
* Contraindication to treatment with fluoropyrimidine, oxaliplatin and irinotecan, including previous unmanageable G3 or greater toxicities, in previous exhibitions.
* Presence of comorbidities that, according to the investigator's assessment, may compromise participant safety
* Prior exposure to the FOLFIRINOX regimen
* Pregnant or lactating women
* Total bilirubin above 1.5mg/dL
* Hepatic transaminases greater than 3 times the upper limit of normality

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Assess response rate after 4 cycles of FOLFIRINOX | 2 years

SECONDARY OUTCOMES:
Progression-free survival | 2 years
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- ICESP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No